CLINICAL TRIAL: NCT06201702
Title: Investigation of the Effect of Pomegranate Supplementation on Symptom Severity in Women With Premenstrual Syndrome: A Randomized Controlled Trial
Brief Title: Effect of Pomegranate Supplementation on Symptom Severity in Women With Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, yasemin hamlacı başkaya, Head of Midwifery Depatment, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 02.01.2024
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Pomegranate; Premenstrual Syndrome
Keywords: premenstrual syndrome; pomegranate; premenstrual symptom; PMS
MeSH Terms: conditions — Premenstrual Syndrome | interventions — pomegranate fruit rind

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the intervention group will first be pre-tested by filling out the data collection tools, and then they will be informed about 3 mL of pomegranate supplementation three times a day for 10 days during 2 menstrual cycles (between 7 days before and 3 days after the estimated onset of menstruation). The test will be repeated at the end of the 2nd month after the intervention
  Interventions: Dietary Supplement: pomegranate extract
- Control group (No Intervention): Participants in the control group will be pre-tested and post-tested after 2 menstrual cycles and at the end of menstrual bleeding. This group will not receive any intervention.

INTERVENTIONS:
Dietary Supplement: pomegranate extract — Drink 2 mL of pomegranate extract three times a day for 10 days during the 3 menstrual cycles (from 7 days before to 3 days after the estimated onset of menstruation).
  Arms: Experimental group

SUMMARY:
Premenstrual syndrome (PMS) is a common disorder among women of reproductive age. About 40% of women report problems with their menstrual cycle. Pomegranate supplementation is one of the practices that may reduce symptoms of premenstrual syndrome (PMS). This study was planned to determine the effect of pomegranate supplementation on the severity of premenstrual syndrome (PMS) symptoms. In the study to be conducted in 2023 with women diagnosed with PMS living in Sakarya province, the individuals to be included in the study will be determined by snowball sampling method and those who meet the inclusion criteria will participate in the study. The researchers will divide the participants into control and intervention groups by using NCSS (statistical software) in a 1:1 ratio using a simple block randomization approach based on CONSORT guidelines. The individuals in the control group will first be administered the PMSÖ (Premenstrual Syndrome Rating Scale) and no intervention will be made. Participants in the intervention group will be informed about 3 mL pomegranate supplementation 13,14 three times a day for 10 days during 2 menstrual cycles (between 7 days before and 3 days after the estimated onset of menstruation). The test will be repeated at the end of the 2nd month post-intervention. Normality of continuous data will be assessed by Kolmogorov-Smirnov test. Data will be expressed as mean ± SD or median and interquartile range (IQR) as appropriate. Variables will be compared between the two intervention and placebo groups using Student's T-test (parametric data) or Mann-Whitney (non-parametric data) or chi-square tests (for qualitative indices). Analyses of changes from pre-intervention to post-intervention within the identified groups will be performed using the Dependent Two Sample t Test (normally distributed parameters) or Wilcoxon signed rank test (non-normally distributed and categorical parameters). All statistical calculations will be performed with SPSS software version 18.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is a common disorder among women of reproductive age. Approximately 40% of women report problems with their menstrual cycle. Nonpharmacologic and pharmacologic treatment methods are used to alleviate symptoms. For mild symptoms, the first line of treatment is nonpharmacologic, while severe symptoms are treated with pharmacologic methods, mainly selective serotonin reuptake inhibitors (SSRIs). Recent data suggest that punica granatum (pomegranate) affects estrogen receptors, as do selective estrogen receptor modulators.

Pomegranate is used in a wide range of applications in complementary medicine. In studies conducted in the field of women's health, it is stated that pomegranate reduces menopausal symptoms, despression symptoms, leads to improvements in PCOS (polycystic syndrome) cases, and is frequently used in the prevention of breast cancers.

Due to the side effects of SSRIs, such as nausea and vomiting, fatigue, skin changes and impaired libido, many patients seek alternative natural treatments to alleviate symptoms. Recent studies in the literature report that menopausal women with PCOS and/or breast cancer are turning to punica granatum (pomegranate) instead of SSRIs.

Pomegranate (scientific name: Punica granatum L.) is a plant with estrogen-like effects used as a traditional medicine to treat hormonal imbalances. This fruit is rich in antioxidants such as polyphenols, tannins and anthocyanins. It also has anti mitogenic and phytoestrogenic effects. It also contains the elements calcium, magnesium, iron, zinc, and there are studies in the literature reporting that pomegranate causes a decrease in PMS symptoms for each element it contains.

Considering the antioxidant, phytoestrogen effects and elemental structure of pomegranate, it is thought to be effective in reducing premenstrual syndrome symptoms.

The overall aim of this study was to determine the effect of 8-week pomegranate supplementation on the severity of PMS symptoms.

ELIGIBILITY:
Inclusion Criteria:

Women who experience PMS complaints (those with a PMSS total score of more than 50%) and who volunteer to participate in the research will be included in our study.

Exclusion Criteria:

* History of acute or chronic illness or history of medication and supplement use
* PMSS total score <50%
* Irregular menstrual cycle
* History of allergy to herbal medicine
* Experiencing any stressful event during the intervention

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — premenstrual syndrome is a female-specific syndrome
Enrollment: 60 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
premenstrual syndrome scale | baseline and at the 8th week
  It is a scale aiming to measure the severity of premenstrual symptoms developed by Gençdoğan in 2006 according to DSM III and DSM IV-R. This scale, which is widely used in Turkey, includes 44 statements that the individual marks by thinking about "being in the period of one week before menstruation". The five-point Likert-type PMSQ consists of 9 subscales (depressed affect, anxiety, fatigue, irritability, depressive thoughts, pain, appetite changes, sleep changes, bloating). The lowest score that can be obtained from the scale is 44 and the highest score is 220. Sub-dimension scores are obtained by summing the items in these dimensions and the total score of the PMSQ is calculated by summing the sub-dimension scores. Those with a PMSQ total score of more than 50% are classified as PMS positive. A higher PMSQ score indicates more severe premenstrual symptoms. Cronbach's alpha (α) = .75 for the original scale

SECONDARY OUTCOMES:
WHO Quality Of Life Bref - WHOQOL-BREF | baseline and at the 8th week
  The WHOQOL-BREF consists of (a) Physical health and well-being (seven items); (b) Psychological health and well-being (six items); (c) Social relationships (three items); and (d) Environment (eight items). Each item has a five-point rating scale from 0-4 (or sometimes 1-5); the higher the item score, the better the person's 'quality of life' in the domain covered by that item.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsen DEMİRHAN KAYACIK, Study Director — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No